CLINICAL TRIAL: NCT01497730
Title: Multi-center, Non-comparative Study of Primary Total Knee Arthroplasty (TKA) Functional Performance
Brief Title: 10003 PRO Current Products
Acronym: 10003
Status: Completed | Type: Observational
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 10003
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Osteoarthritis
Keywords: Arthroplasty, Replacement, Knee,
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- CR FB: Subjects receiving a Cruciate Retaining Fixed Bearing implant configuration
  Interventions: Device: Total Knee Replacement
- PS FB: Subjects Receiving a Posterior Stabilized Fixed Bearing implant configuration
  Interventions: Device: Total Knee Replacement
- CR RP: Subjects receiving a Cruciate Retaining Rotating Platform implant configuration
  Interventions: Device: Total Knee Replacement
- PS RP: Subjects receiving a Posterior Stabilized Rotating Platform implant configuration
  Interventions: Device: Total Knee Replacement

INTERVENTIONS:
Device: Total Knee Replacement — Subjects will receive one of the following total knee implants:
  PFC Sigma Fixed Bearing (FB) cruciate retaining (CR), posterior stabilized (PS) or Rotating Platform CR or PS devices. LCS Rotating platform or PS devices. Triathlon CR, PS or mobile bearing devices. NexGen CR, LPS, LPS Flex FB PS, LPS Flex Mobile bearing, or LPS Mobile bearing devices.

SUMMARY:
This post-marketing investigation will evaluate the functional knee performance of Subjects who have undergone primary total knee arthroplasty (TKA). Data from Subjects who receive one of four contemporary knee configurations from different manufacturers will be pooled to establish a contemporary dataset.

The primary objective of this study is to evaluate the functional performance as measured by the activities of daily living (ADL) sub-score of the Knee Osteoarthritis Outcomes Score (KOOS) patient-reported outcome (PRO) questionnaire of primary TKA at minimum one year post-operation. This will be carried out for all four implant configurations. The final endpoint is a 2-year evaluation.

DETAILED DESCRIPTION:
The study is designed as a prospective, single arm stratified, multi-center investigation.

Approximately 20 study sites, worldwide, will enroll 840 patients (840 knees). Each study site is expected to enroll approximately 42 patients (42 knees). Cohort reallocation is permitted. There will be no control group. Eight hundred forty (840) Subjects will be stratified into 4 subgroups of 210: fixed bearing cruciate retaining (FB CR), fixed bearing posterior stabilized (FB PS), rotating platform cruciate retaining (RP CR), and rotating platform posterior stabilized (RP PS).

Treatment assignment in this study is not randomized. Each site will only enroll patients in one of the four knee configuration sub-groups most commonly used as their standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and between the ages of 22 and 80 years, inclusive.
* Subject was diagnosed with NIDJD.
* Subject is a suitable candidate for cemented primary TKA using the devices described in this CIP with either a resurfaced or non-resurfaced patellae.
* Subject's TKA device was one of the total knee prostheses described under Interventions.
* Subject is currently not bedridden.
* Subject has given voluntary, written informed consent to participate in this clinical investigation, is willing and able to perform all study procedures and follow-up visits and has authorized the transfer of his/her information to DePuy.
* Subject, in the opinion of the Clinical Investigator, is able to understand this clinical investigation and co-operate with investigational procedures.
* Subject must be comfortable with speaking, reading, and understanding questions and providing responses in English.
* The devices specified in this CIP were implanted.

Exclusion Criteria:

* The Subject is a woman who is pregnant or lactating.
* Contralateral knee has already been enrolled in this study.
* Subject had a contralateral amputation.
* Previous partial knee replacement (unicompartmental, bicompartmental or patellofemoral joint replacement), patellectomy, high tibial osteotomy or primary TKA in affected knee.
* Subject is currently experiencing radicular pain from the spine.
* Subject has participated in an IDE/IND clinical investigation with an investigational product in the last three months.
* Subject is currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
* Subject is a known drug or alcohol abuser or has a psychological disorder that could affect their ability to complete patient reported questionnaires.
* Subject was diagnosed with fibromyalgia that is currently being treated with prescription medication.
* Subject has significant neurological or musculoskeletal disorders or disease that may adversely affect gait or weight bearing (e.g. muscular dystrophy, multiple sclerosis, Charcot disease).
* Subject is suffering from inflammatory arthritis (e.g. rheumatoid arthritis, juvenile rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus, etc.).
* Subject is not comfortable with speaking, reading, and understanding questions and providing responses in an available translated language for the PROs in the CIP.
* Subject has a medical condition with less than 2 years of life expectancy.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female Subjects with Non-inflammatory Degenerative Joint Disease (NIDJD) who require primary TKA with one of several designated knee systems currently on the market and are aged 22 to 80 years, inclusive.
Sampling Method: Non-Probability Sample
Enrollment: 842 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) activities of daily living (ADL) sub-score | up to one year
  The primary endpoint will be measuerd before surgery and out to a minimum of 1 year after surgery. The KOOS is a patient self-administered questionnaire that consists of 42 questions. The KOOS consists of 5 subscales; pain, other symptoms, activities of daily living (ADL), sport and recreational function and knee-related quality of life. Each question has 5 Likert-like response options. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.

SECONDARY OUTCOMES:
Evaluate the psychometric properties of PKIP | Pre-op (-90 to -1 days before surgery), < 1 year (1 to 303 days), minimum 1 year (304 to 668 days), minimum 2 year (669 to 1763 days)
  The Pre and Post-Surgical Patient's Knee Implant Performance (PKIP) questionnaire is a patient self-administered questionnaire that consists of 25 questions relating to the patient's awareness of their knee. Questions include the patient's self-confidence about the current status of their knee performance, stability, and overall satisfaction. Each question has a 5, 6 or 10 Likert- like response option.
Evaluate the longitudinal functional performance of primary TKA | < 1 year (1 to 303 days), minimum 1 year (304 to 668 days), minimum 2 year (669 to 1763 days)
Evaluate Incidence of Anterior Knee Pain | Pre-op (-90 to -1 days before surgery), < 1 year (1 to 303 days), minimum 1 year (304 to 668 days), minimum 2 year (669 to 1763 days)
Evaluate incidence of asymptomatic and symptomatic crepitus | Pre-op (-90 to -1 days before surgery), < 1 year (1 to 303 days), minimum 1 year (304 to 668 days), minimum 2 year (669 to 1763 days)
Evaluate patients functional performance for PS knees, CR knees, FB knees, and RP knees | < 1 year (1 to 303 days), minimum 1 year (304 to 668 days), minimum 2 year (669 to 1763 days)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad S. Ismail, MS, CCRP, Study Director — DePuy Orthopaedics
Locations (22):
- United States (11):
  - Orthopaedic Specialty Institute, Orange, California
  - UCSD Medical Center, San Diego, California
  - Orthopaedic Center of the Rockies, Fort Collins, Colorado
  - Heekin Institute for Orthopedic Research, Jacksonville, Florida
  - The Arthroplasty Foundation, Louisville, Kentucky
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Hip and Knee Research of Nevada, Las Vegas, Nevada
  - Dartmouth Medical School/Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cardinal Orthopaedic Institute, Columbus, Ohio
  - Anderson Orthopaedic Research Institute, Alexandria, Virginia
  - Swedish Orthopedic Institute, Seattle, Washington
- Australia (4):
  - Hornsby Ku-ring-gai Hospital, Hornsby, New South Wales
  - Wakefield Orthopedic Clinic, Adelaide, South Australia
  - Freemantle Hospital, Crawley, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Ascot Hospital, Auckland, New Zealand
- United Kingdom (6):
  - Queen Margaret Hospital, Dunfermline, Fife
  - The Royal Surrey County Hospital, Guildford, Surrey
  - Princess Alexandra Hospital, Harlow
  - University Hospital Llandough, Llandough
  - James Cook University Hospital, Middlesbrough
  - Clifton Park NHS Treatment Centre, York

REFERENCES:
- [Derived] Hamilton WG, Brenkel IJ, Barnett SL, Allen PW, Dwyer KA, Lesko JP, Kantor SR, Clatworthy MG. Comparison of Existing and New Total Knee Arthroplasty Implant Systems From the Same Manufacturer: A Prospective, Multicenter Study. J Am Acad Orthop Surg Glob Res Rev. 2021 Dec 15;5(12):e21.00136. doi: 10.5435/JAAOSGlobal-D-21-00136. PMID 34908561